CLINICAL TRIAL: NCT01788644
Title: Nurture: Early Child Care and Risk of Obesity
Brief Title: Early Child Care and Risk of Obesity
Acronym: Nurture
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00036242
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Child Adiposity
Keywords: Child adiposity; Infancy; Motor activity; Feeding behavior; Sleep; Stress, Physiological
MeSH Terms: conditions — Motor Activity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, fecal
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment (observational study)

SUMMARY:
The purpose of this study is to examine risk factors associated with infant growth and the development of obesity in the first year of life. The investigators plan to establish a racially and ethnically diverse southern cohort of 800 mother/infant dyads, followed regularly from birth to 12 months of age. The cohort will be residents of Durham, North Carolina (NC) and the immediate surrounding area. The proposed longitudinal study will examine factors contributing to the development of obesity, including dietary behaviors, physical activity and inactivity, stress, and sleep duration and quality. Frequent in-home assessments throughout infancy and contact with other care providers will help pinpoint exactly when children begin to gain weight excessively and will identify risk factors related to energy intake, energy expenditure, stress, and sleep associated with obesity.

ELIGIBILITY:
Inclusion Criteria:

* mother over 18
* in 2nd or 3rd trimester of pregnancy with singleton
* speak and read English
* planning to stay in area for the first year of baby's life

Exclusion Criteria:

* baby born with conditions that may affect weight, feeding or motor activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mothers/infant dyads in the Durham, NC area
Sampling Method: Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in child adiposity | birth - 12 months
  In-person assessments of infant weight, length, and skinfold thicknesses at birth, 3, 6, 9, and 12 months of age

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Benjamin Neelon SE, Ostbye T, Bennett GG, Kravitz RM, Clancy SM, Stroo M, Iversen E, Hoyo C. Cohort profile for the Nurture Observational Study examining associations of multiple caregivers on infant growth in the Southeastern USA. BMJ Open. 2017 Feb 8;7(2):e013939. doi: 10.1136/bmjopen-2016-013939. PMID 28179416
- [Result] Costa S, Adams J, Gonzalez-Nahm S, Benjamin Neelon SE. Childcare in Infancy and Later Obesity: a Narrative Review of Longitudinal Studies. Curr Pediatr Rep. 2017;5(3):118-131. doi: 10.1007/s40124-017-0134-7. Epub 2017 Jun 15. PMID 28845369
- [Result] Khatiwada A, Shoaibi A, Neelon B, Emond JA, Benjamin-Neelon SE. Household chaos during infancy and infant weight status at 12 months. Pediatr Obes. 2018 Oct;13(10):607-613. doi: 10.1111/ijpo.12395. Epub 2018 Jul 17. PMID 30019385
- [Result] Hesketh KR, Evenson KR, Stroo M, Clancy SM, Ostbye T, Benjamin-Neelon SE. Physical activity and sedentary behavior during pregnancy and postpartum, measured using hip and wrist-worn accelerometers. Prev Med Rep. 2018 Apr 19;10:337-345. doi: 10.1016/j.pmedr.2018.04.012. eCollection 2018 Jun. PMID 29868389
- [Derived] Emond JA, O'Malley AJ, Neelon B, Kravitz RM, Ostbye T, Benjamin-Neelon SE. Associations between daily screen time and sleep in a racially and socioeconomically diverse sample of US infants: a prospective cohort study. BMJ Open. 2021 Jun 24;11(6):e044525. doi: 10.1136/bmjopen-2020-044525. PMID 34168024